CLINICAL TRIAL: NCT06347666
Title: Equity-focused Implementation of Caregiver Coaching for Unhoused Children At-risk for Developmental Delay
Brief Title: Coaching in Early Development Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23082905
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: One group will receive the caregiver coaching intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver Coaching (Experimental): In this arm, participants receive a caregiver coaching intervention. In the intervention, a speech language pathologist offers strategies to support child development.
  Interventions: Behavioral: Caregiver coaching

INTERVENTIONS:
Behavioral: Caregiver coaching — Speech language pathologists will meet with caregivers to talk through strategies to promote child development.

SUMMARY:
Among young children, homelessness is an independent predictor of child developmental delay and disability, and children experiencing homelessness (CEH) are 2-4x more likely to demonstrate developmental delays compared to housed children. The purpose of this project is to evaluate an evidence-based model of caregiver coaching for CEH that screen positive for developmental delay. The investigators will also evaluate the societal costs of the program, its preliminary efficacy, and the acceptability among caregivers and shelter staff.

DETAILED DESCRIPTION:
Over 2.5 million children experience homelessness (CEH) in a given year and housing intersects with inequities due to race and disability. Among young children, homelessness is an independent predictor of child developmental delay and disability, and CEH are 2-4x more likely to demonstrate developmental delays compared to housed children. Caregiver coaching is an evidence-based and effective behavioral therapy method to support child development and has been recommended by the American Academy of Pediatrics for adoption across all early intervention (EI) systems. EI is mandated by states under the Individuals with Disabilities Education Act (IDEA) Part C and provides behavioral therapy for all children ages 0-3 years that show developmental delay. Within EI, caregiver coaching is delivered is delivered in families' homes, and therefore has limited evaluation of implementation in shelters. In ongoing pilot work, in collaboration with shelter-based primary care, 70% of CEH screened positive for developmental delay, yet no child received caregiver coaching through EI. Therefore, the objective of this proposal is to use a Type II Hybrid Trial to investigate how implementation strategies influence uptake of shelter-based caregiver coaching and subsequent child outcomes. The proposed study will use implementation research as a guide to evaluate our team's implementation of caregiver coaching from an equity lens among a population that consistently lacks access to evidence-based interventions to improve children's developmental trajectories. Specifically, the investigators will 1) Evaluate implementation of a 12-week shelter-based caregiver coaching intervention on caregiver attendance and fidelity (i.e., adherence) among CEH with delay ages compared to statewide equity metrics; 2) Evaluate the societal costs of implementing a 12-week shelter-based caregiver coaching intervention; 3) Investigate facilitators and barriers related to attendance and fidelity of a 12-week coaching intervention among caregivers of CEH and shelter staff; 4) Explore the efficacy of the 12-week coaching intervention on caregiver and child outcomes. While disparities in access to evidence-based developmental care for CEH is documented, the investigators will identify how strategies that promote equity in access result in caregiver uptake and costs. By evaluating stakeholder feedback of an evidence-based intervention not yet tested in shelters, the investigators can integrate changes to the model for future trials. The impact will be on prioritizing ways to promote uptake of tailored developmental interventions for children most in need, ultimately contributing to evidence to share with families, shelters, and policymakers to create sustainable models of care.

ELIGIBILITY:
Inclusion Criteria:

* Children must be unhoused or experience housing instability and screen positive for developmental delay

Exclusion Criteria:

* Children are excluded if they are receiving more than 1 hour/week of early intervention

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Parenting Sense of Competence Scale | baseline and post-12 week intervention
  Self-report of satisfaction and efficacy associated with parenting. Higher scores mean that a respondent has higher parenting sense of competence. Scores range from 6-102.
Parenting Stress Scale | baseline and post-12 week intervention
  Self-report of stressors associated with parenting. Higher scores mean higher parenting stress and scores range from 18-90.

SECONDARY OUTCOMES:
Mullen Scales of Early Learning | baseline and post-12 week intervention
  Behavioral assessment of overall child development. Scores are presented as standard scores with a mean of 50 and a standard deviation of 10. Higher standard scores mean increased overall development.
Maternal Behavior Responsivity Scale | baseline and post-12 week intervention
  Observational assessment of maternal responsivity. Higher scores mean increased maternal responsivity. Scores range from 5-25.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Little, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the small sample size of the study, leading to potential privacy concerns.